CLINICAL TRIAL: NCT07227363
Title: Symptoms of Polycystic Ovarian Syndrome Ameliorated by Keto-Adaptation Pilot
Acronym: (SPARK-Pilot)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Madison Kackley, Assistant Professor, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2023H0368
Record Dates: First submitted 2025-11-06; First posted 2025-11-12 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: PCOS (Polycystic Ovary Syndrome)
Keywords: Ketogenic Diet; Exogenous Ketones; Nutritional Ketosis; Reproductive Hormones; Ovarian Function; Women's Health; Metabolic Health; PCOS
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Diet, Ketogenic

STUDY DESIGN:
Masking Description: This is a pilot feasibility study; therefore, no masking will be implemented. Participants and investigators will be aware of group assignments due to the distinct nature of the dietary and supplement interventions. The study is designed as an open-label trial to evaluate adherence, feasibility, and physiological responses to each intervention before planning a larger randomized, controlled study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ketogenic Diet (KD) (Experimental): Participants in this arm will follow a well-formulated ketogenic diet designed to achieve and maintain nutritional ketosis (β-hydroxybutyrate ≥0.5 mmol/L). The diet will include non-starchy vegetables as the primary carbohydrate source (20-50 g/day), moderate protein (1.2-1.6 g/kg/day), and sufficient fat for energy and satiety. All meals and snacks will be provided for the first 2 weeks, followed by self-guided adherence with support from the study dietitian and educational resources. Daily fingerstick ketone and glucose levels will be monitored using KetoMojo.
  Interventions: Other: Ketogenic diet
- Mixed Diet + Exogenous Ketone Supplement (Active Comparator): Participants in this arm will follow a balanced, mixed diet aligned with USDA macronutrient recommendations while consuming an exogenous ketone supplement throughout the 12-week intervention. The supplement is designed to raise circulating β-hydroxybutyrate to nutritional ketosis levels without carbohydrate restriction. As with the KD arm, all meals and snacks will be provided for the first 2 weeks, followed by self-guided adherence with ongoing dietitian support.
  Interventions: Dietary Supplement: Exogenous Ketone Supplement

INTERVENTIONS:
Other: Ketogenic diet — A well-formulated ketogenic diet designed to achieve nutritional ketosis (β-hydroxybutyrate ≥0.5 mmol/L). The diet emphasizes non-starchy vegetables as the primary carbohydrate source (20-50 g/day), moderate protein intake (1.2-1.6 g/kg/day), and sufficient dietary fat for energy and satiety. All meals and snacks will be provided during the initial two weeks, followed by a self-guided phase with ongoing dietitian support and education materials. Participants will monitor daily fasting ketones and glucose using a handheld analyzer (KetoMojo).
  Arms: Ketogenic Diet (KD)
Dietary Supplement: Exogenous Ketone Supplement — A dietary supplement containing a ketone ester designed to elevate circulating β-hydroxybutyrate concentrations to nutritional ketosis levels without carbohydrate restriction. Participants will consume the supplement throughout the 12-week intervention while following a balanced, mixed diet consistent with USDA dietary guidelines.
  Arms: Mixed Diet + Exogenous Ketone Supplement

SUMMARY:
The SPARK- Pilot study (Symptoms of PCOS Ameliorated by Responses to Keto-adaptation) is a 12-week clinical trial at The Ohio State University designed to explore how different ways of achieving ketosis may improve reproductive and metabolic health in women with Polycystic Ovary Syndrome (PCOS).

Participants will be randomly assigned to one of two groups:

* A ketogenic diet group, following a low-carbohydrate, nutrient-dense meal plan.
* A mixed diet plus ketone supplement group, following general dietary guidelines while taking an exogenous ketone supplement.

The study will measure whether these approaches help restore regular ovulation and improve hormone balance, metabolism, and overall well-being. Optional imaging using MRI will also examine heart and ovarian health.

This pilot study will help researchers understand if ketogenic nutrition strategies are a safe, effective way to support menstrual regularity and reduce PCOS-related symptoms, providing groundwork for larger clinical trials.

DETAILED DESCRIPTION:
The SPARK study (Symptoms of PCOS Ameliorated by Responses to Keto-adaptation) is a 12-week randomized, two-arm intervention examining how nutritional ketosis influences ovulatory and metabolic outcomes in women with Polycystic Ovary Syndrome (PCOS).

PCOS is a common endocrine disorder that affects hormone balance, menstrual function, and metabolism. Current treatments often address single symptoms but rarely provide comprehensive improvement. Ketogenic dietary interventions have shown promise for improving insulin sensitivity, hormone profiles, and body composition; however, few studies have evaluated their direct impact on ovulation.

In this pilot trial, 40 women aged 18-40 years with diagnosed PCOS will be randomized to one of two groups:

Ketogenic Diet (KD): Participants will follow a low-carbohydrate, high-fat, moderate-protein diet designed to achieve and maintain nutritional ketosis (β-hydroxybutyrate ≥0.5 mmol/L).

Mixed Diet + Exogenous Ketone Supplement: Participants will consume a balanced diet aligned with USDA macronutrient recommendations and receive a ketone ester supplement.

Primary outcomes include changes in ovulatory status, assessed through hormonal markers, ovulation prediction tests, and continuous basal body temperature monitoring (OvuSense). Secondary outcomes include changes in reproductive hormones (progesterone, estrogen, LH, FSH), metabolic and lipid markers, and exploratory imaging of cardiovascular function and ovarian morphology via MRI.

This study will provide feasibility and preliminary efficacy data to inform a future large-scale clinical trial evaluating ketogenic strategies for improving menstrual regularity and overall health in women with PCOS.

ELIGIBILITY:
Inclusion Criteria:

* Female participants aged 18-40 years.
* Clinical diagnosis of Polycystic Ovary Syndrome (PCOS) according to Rotterdam criteria (presence of at least two of the following: oligo- or anovulation, clinical or biochemical signs of hyperandrogenism, and/or polycystic ovaries on ultrasound).
* Willingness and ability to comply with all study procedures, including fasting (>10 hours; water only), avoidance of alcohol (>24 hours), and abstaining from exercise (>24 hours) prior to each test visit.
* Willing to maintain current diet, exercise, medication, and supplement habits throughout the study.
* Body mass index (BMI) ≥18 kg/m².
* Access to a smartphone, computer, or tablet for digital tracking and study communication.

Exclusion Criteria:

* Current adherence to a low-carbohydrate diet (<30% of total energy from carbohydrates).
* Non-PCOS etiologies of anovulation (e.g., menopause, oophorectomy, or other reproductive disorders).
* History of type 1 diabetes or uncontrolled type 2 diabetes.
* Weight loss ≥10% of body weight within the previous 6 months.
* Pregnancy or breastfeeding.
* Use of hormonal contraception or medications known to alter reproductive hormones within 3 months prior to enrollment.
* Active eating disorder or medical condition that could interfere with dietary intervention.
* Any condition that, in the opinion of the Investigator, could interfere with participation, data integrity, or safety.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — This study enrolls biological females aged 18-40 years who have been clinically diagnosed with PCOS. Because the primary outcomes involve menstrual cyclicity, ovulatory function, and reproductive hormone regulation, eligibility is limited to individuals assigned female at birth. Self-identified women meeting these criteria are eligible to participate, regardless of gender identity, provided they have intact ovarian function and are not pregnant or breastfeeding.
Enrollment: 40 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in Ovulatory Status | Baseline to 12 weeks
  To evaluate whether ketogenic dietary intervention or exogenous ketone supplementation restores ovulatory function in women with Polycystic Ovary Syndrome (PCOS). Ovulatory status will be assessed using a combination of validated measures, including basal body temperature monitoring via BBT, urinary luteinizing hormone (LH) surge detection using ovulation predictor kits, and serum progesterone levels. Participants will be classified as ovulatory or anovulatory based on hormonal and temperature cycle confirmation.

SECONDARY OUTCOMES:
Change in Serum Progesterone Concentration (ng/mL) | Baseline to 12 weeks
  To determine the effects of ketogenic diet and exogenous ketone supplementation on circulating reproductive hormone concentrations. Serum progesterone will be analyzed using standard immunoassay techniques (Quest Diagnostics panels and/or validated ELISA assays). Hormonal changes will be compared between baseline and post-intervention to assess improvements in reproductive axis regulation.
Change in Serum Estradiol Concentration (pg/mL) | Baseline to 12 weeks
  To determine the effects of ketogenic diet and exogenous ketone supplementation on circulating reproductive hormone concentrations. Serum estradiol will be analyzed using commercially available immunoassay kits (Quest Diagnostics panels and/or validated ELISA assays). Hormonal changes will be compared between baseline and post-intervention to assess improvements in reproductive axis regulation.
Change in Serum Luteinizing Hormone Concentration (mIU/mL) | Baseline to 12 weeks
  To determine the effects of ketogenic diet and exogenous ketone supplementation on circulating reproductive hormone concentrations. Serum luteinizing hormone (LH) will be analyzed using standard immunoassay techniques (Quest Diagnostics panels and/or validated ELISA assays). Hormonal changes will be compared between baseline and post-intervention to assess improvements in reproductive axis regulation.
Change in Serum Follicle Stimulating Hormone Concentrations (mIU/mL) | Baseline to 12 weeks
  To determine the effects of ketogenic diet and exogenous ketone supplementation on circulating reproductive hormone concentrations. Serum follicle-stimulating hormone (FSH) will be analyzed using standard immunoassay techniques (Quest Diagnostics panels and/or validated ELISA assays). Hormonal changes will be compared between baseline and post-intervention to assess improvements in reproductive axis regulation.
Change in Daily Fasting BHB (mmol/L) | Baseline to 12 weeks (Daily)
  To assess changes in metabolic parameters including fasting β-hydroxybutyrate (BHB). Capillary ketones will be measured daily using KetoMojo handheld monitors.
Change in Daily Fasting Glucose (mg/dL) | Baseline to 12 weeks (Daily)
  To assess changes in metabolic parameters including fasting glucose. Capillary glucose will be measured daily using KetoMojo handheld monitors.
Change in Serum Insulin Concentration (µIU/mL) | Baseline to 12 weeks
  To assess the effect of ketogenic diet and exogenous ketone supplementation on fasting insulin levels. Serum insulin will be measured at laboratory visits via immunoassay (Quest Diagnostics or validated ELISA). Mean change from baseline will be compared across groups.
Change in Serum Total Cholesterol Concentration (mg/dL) | Baseline to 12 weeks
  To assess changes in fasting serum total cholesterol in response to ketogenic diet and exogenous ketone supplementation. Blood samples will be collected biweekly and analyzed using standard clinical chemistry methods (Quest Diagnostics). Mean change from baseline to 12 weeks will be reported.
Change in Serum Triglyceride Concentration (mg/dL) | Baseline to 12 weeks
  To determine the effect of ketogenic diet and exogenous ketone supplementation on fasting triglyceride concentrations. Serum triglycerides will be measured via standard lipid panel. Mean change from baseline to 12 weeks will be compared across groups.
Change in Serum LDL Cholesterol Concentration (mg/dL) | Baseline to 12 weeks
  To assess the effect of ketogenic diet and exogenous ketone supplementation on fasting low-density lipoprotein (LDL) cholesterol. Serum LDL will be measured via standard lipid panel (Quest Diagnostics). Mean change from baseline to post-intervention will be reported.
Change in Serum HDL Cholesterol Concentration (mg/dL) | Baseline to 12 weeks
  To evaluate changes in fasting high-density lipoprotein (HDL) cholesterol following ketogenic diet or exogenous ketone supplementation. Serum HDL will be analyzed by clinical chemistry methods. Mean change from baseline to 12 weeks will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Madison Kackley, PhD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided
This is an early-stage pilot study focused on feasibility and exploratory outcomes. At this stage, individual participant data (IPD) will not be publicly shared until all analyses are complete and findings are published. De-identified aggregate data may be shared upon reasonable request following publication, in accordance with institutional and IRB policies. If a larger, follow-up trial is initiated, a formal data-sharing plan will be developed to align with NIH and ICMJE requirements.

DOCUMENTS (1):
  • Study Protocol (2025-10-14): https://cdn.clinicaltrials.gov/large-docs/63/NCT07227363/Prot_000.pdf